CLINICAL TRIAL: NCT02390154
Title: A Phase I, Single Center, Open-label, Non-randomized, Non-placebo-controlled Study to Investigate the Metabolism, Excretion Pattern, Mass Balance, Safety, Tolerability and Pharmacokinetics of Orally Administered [14C]-Roniciclib (BAY 1000394) in Patients With Solid Tumors
Brief Title: Roniciclib Mass Balance Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15022; 2014-002797-37 (EudraCT Number)
Record Dates: First submitted 2015-03-11; First posted 2015-03-17 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — roniciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Open label non-randomized non-controlled mass balance study in Cycle 1
  Interventions: Drug: roniciclib (BAY 1000394)
- Arm 2 (Experimental): Open label non-randomized non controlled multiple dose study in Cycle 2 and subsequent cycles
  Interventions: Drug: roniciclib (BAY 1000394)

INTERVENTIONS:
Drug: roniciclib (BAY 1000394) — Single dose , 2.5 mg roniciclib spiked with 5.0 MBq of [14C] roniciclib solution
  Arms: Arm 1
Drug: roniciclib (BAY 1000394) — 5 mg roniciclib tablet , Multiple dose, twice a day (bid), on a 3-days on/4-days off regimen in cycles of 21 days
  Arms: Arm 2

SUMMARY:
The purpose of this trial is to investigate the fate of the roniciclib (study drug) in the body in a so called mass-balance study. This means to investigate how the study drug is absorbed, distributed, broken down (metabolized) and removed (excreted or eliminated) from the body.

ELIGIBILITY:
Inclusion Criteria:

* - Male or female subjects aged ≥18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2
* Subjects with advanced, histologically or cytologically confirmed solid tumors, refractory to any standard therapy, have no standard therapy available, or subjects must have actively refused any treatment which would be regarded standard, and / or if in the judgment of the investigator, experimental treatment is clinically and ethically acceptable
* Adequate bone marrow, liver, and renal functions as assessed by laboratory requirements to be conducted within 14 days prior to the first dose of study drug:

Exclusion Criteria:

* Previous deep vein thrombosis (within the last 6 months), arterial thrombotic events (including strokes), or pulmonary embolism
* History of cardiac disease: congestive heart failure New York Heart Association (NYHA) class III or IV, angina (within past 6 months prior to study entry), myocardial infarction, or cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted)
* Anticancer chemotherapy or immunotherapy within 4 weeks of study entry. Mitomycin C or nitrosoureas should not be given within 6 weeks of study entry. Accepted exemptions are bisphosphonates, luteinising hormone releasing hormone (LHRH) agonists for prostate cancer, and mitotane for adrenal carcinoma.
* Radiotherapy within 3 weeks prior to the first dose of study drug. Palliative radiotherapy will be allowed
* Intake of strong CYP3A4 inhibitors (e.g., boceprevir, clarithromycin, conivaptan, indinavir, itraconazole, ketoconazole, lopinavir/ritonavir, mibefradil (withdrawn in the US), nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telaprevir, telithromycin and voriconazole) and strong CYP3A4 inducers (e.g., carbamazepine, phenytoin , rifampin and St. John's Wort)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-04; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Amount of Roniciclib in urine as percentage of the dose of total radioactivity. | Up to 336 hours
Amount of Roniciclib in feces as percentage of the dose of total radioactivity. | Up to 336 hours
Amount of Roniciclib in vomit as percentage of the dose of total radioactivity | Up to 336 hours
Cmaxof roniciclib in plasma | up to 336 hours
AUC(0-tlast) of roniciclib in plasma | up to 336 hours
AUC of roniciclib in plasma | up to 336 hours
Cmax of total radioactivity in whole blood and plasma | up to 336 hours
AUC(0-tlast) of total radioactivity in whole blood and plasma | Up to 336 hours
AUC of total radioactivity in whole blood and plasma | up to 336 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- PRA Magyarorszag Kft. Fazis I-es Klin.Farmakol. Vizsgalohely, Budapest, Hungary